CLINICAL TRIAL: NCT00175942
Title: Indicators of Coagulation Activation and Inflammation Contributing to Ventricular Fibrillation Complicating Acute Myocardial Infarction
Brief Title: Risk Indicators in Patients With Ventricular Fibrillation During Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Other Study IDs: 0229.3
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-05

CONDITIONS: Acute Myocardial Infarction; Sudden Cardiac Death
Keywords: acute myocardial infarction; ventricular fibrillation; coagulation; inflammation
MeSH Terms: conditions — Death, Sudden, Cardiac; Ventricular Fibrillation; Thrombosis; Inflammation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Sudden cardiac death is in most cases triggered by ischemia-related ventricular tachyarrhythmias and accounts for 50% of deaths from cardiovascular disease in developed countries. Chronic elevation of indicators of coagulation activation has been found in patients with coronary heart disease , but a role of coagulation activation and proinflammatory state as a potential risk factor for ventricular fibrillation (VF) during acute myocardial infarction has not been investigated.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) is in most cases triggered by ischemia-related ventricular arrhythmias and is responsible for 50% of the mortality from cardiovascular disease in developed countries (1). Chronic elevation of indicators of coagulation activation and inflammation has been found in patients with coronary heart disease and may contribute to vasculatory disorders probably contributing to the development of arrhythmogenesis. However, the role of coagulation activation as a potential risk factor for ventricular fibrillation during acute myocardial infarction has not been investigated yet.

ELIGIBILITY:
Inclusion Criteria:

ST-elevation myocardial infarction ventricular fibrillation during acute MI

Exclusion Criteria:

NSTEMI coagulation disorders, e.g.intake of coumadin

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2003-02

CONTACTS AND LOCATIONS:
Overall Officials: Carl E. Dempfle, Prof.Dr., Principal Investigator — University Hospital of Mannheim, University of Heidelberg
Locations (1):
- University Hospital of Mannheim, University of Heidelberg, Mannheim, Germany